CLINICAL TRIAL: NCT00643890
Title: Phase 2 Safety and Efficacy Study Evaluating Glutamic Acid Decarboxylase Gene Transfer to Subthalamic Nuclei in Subjects With Advanced Parkinson's Disease
Brief Title: Study of AAV-GAD Gene Transfer Into the Subthalamic Nucleus for Parkinson's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to financial reasons
Sponsor: Neurologix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRGX-GAD-02
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Parkinson's Disease
Keywords: Keywords:; Parkinson's disease; Gene transfer; Gene therapy; Subthalamic nucleus; Adeno-associated virus; Study placed in the following topic categories:; Ganglion Cysts; Movement Disorders; Parkinson Disease; Basal Ganglia Diseases; Central Nervous System Diseases; Parkinsonian Disorders; Neurodegenerative Diseases; Brain Diseases; Additional relevant MeSH terms:; Nervous System Diseases
MeSH Terms: conditions — Parkinson Disease; Ganglion Cysts; Movement Disorders; Basal Ganglia Diseases; Central Nervous System Diseases; Parkinsonian Disorders; Neurodegenerative Diseases; Brain Diseases; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: Bilateral surgical infusion of AAV-GAD into the subthalamic nucleus — One-time bilateral administration of rAAV-GAD at 1X10^12 vector genomes in 35 uL.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of AAV-GAD gene transfer into the subthalamic nucleus (STN) region of the brain. This study involves the treatment of subjects with medically refractory Parkinson's disease (PD). The gene transfer product, a disabled virus with a gene called GAD, will be infused into the STN bilaterally using stereotactic surgical techniques. The overall goal of this approach is to normalize the activity of the STN and reduce the motor symptoms of PD.

Because the change in UPDRS demonstrated a positive outcome, the sham surgery subjects from the blinded portion of the study will be invited to crossover into the Open-label Arm portion of the study. The Open-label Arm will further evaluate the safety and efficacy of AAV-GAD gene transfer into the subthalamic nucleus (STN) region of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Duration of disease for at least 5 years
* Levodopa responsiveness for at least 12 months
* UPDRS Part 3 score ≥ 25 or more in "off" state

Exclusion Criteria:

* Past history of brain surgery for PD
* Beck Depression Inventory Score ≥ 20
* Any history of cerebral insult or central nervous system infection
* Cognitive impairment score < 130 on the Mattis Dementia Rating Scale
* Focal neurological deficits
* Evidence of significant medical or psychiatric disorders
* Secondary Parkinsonism
* Atypical Parkinson's disease
* History of substance abuse

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluate a change in UPDRS scores

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health Systems - Franklin Pointe Medical, Southfield, Michigan
  - University of Rochester, Rochester, New York
  - Wake Forest University Health Science Center, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] Kaplitt MG, Feigin A, Tang C, Fitzsimons HL, Mattis P, Lawlor PA, Bland RJ, Young D, Strybing K, Eidelberg D, During MJ. Safety and tolerability of gene therapy with an adeno-associated virus (AAV) borne GAD gene for Parkinson's disease: an open label, phase I trial. Lancet. 2007 Jun 23;369(9579):2097-105. doi: 10.1016/S0140-6736(07)60982-9. PMID 17586305
- [Background] Feigin A, Kaplitt MG, Tang C, Lin T, Mattis P, Dhawan V, During MJ, Eidelberg D. Modulation of metabolic brain networks after subthalamic gene therapy for Parkinson's disease. Proc Natl Acad Sci U S A. 2007 Dec 4;104(49):19559-64. doi: 10.1073/pnas.0706006104. Epub 2007 Nov 27. PMID 18042721
- [Result] LeWitt PA, Rezai AR, Leehey MA, Ojemann SG, Flaherty AW, Eskandar EN, Kostyk SK, Thomas K, Sarkar A, Siddiqui MS, Tatter SB, Schwalb JM, Poston KL, Henderson JM, Kurlan RM, Richard IH, Van Meter L, Sapan CV, During MJ, Kaplitt MG, Feigin A. AAV2-GAD gene therapy for advanced Parkinson's disease: a double-blind, sham-surgery controlled, randomised trial. Lancet Neurol. 2011 Apr;10(4):309-19. doi: 10.1016/S1474-4422(11)70039-4. PMID 21419704
- [Derived] Niethammer M, Tang CC, LeWitt PA, Rezai AR, Leehey MA, Ojemann SG, Flaherty AW, Eskandar EN, Kostyk SK, Sarkar A, Siddiqui MS, Tatter SB, Schwalb JM, Poston KL, Henderson JM, Kurlan RM, Richard IH, Sapan CV, Eidelberg D, During MJ, Kaplitt MG, Feigin A. Long-term follow-up of a randomized AAV2-GAD gene therapy trial for Parkinson's disease. JCI Insight. 2017 Apr 6;2(7):e90133. doi: 10.1172/jci.insight.90133. PMID 28405611